CLINICAL TRIAL: NCT07033312
Title: Therapeutic Effect of Combined Treatment of Oral Nutritional Supplement Based on Hyaluronic Acid With Hyaluronic Acid Intra-articular Injection on Symptomatic Knee Osteoarthritis
Brief Title: Therapeutic Effect of Oral Hyaluronic Acid on Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SF22377A
Record Dates: First submitted 2025-06-01; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: both the patients and the investigators were blinded to the agent patients took
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oral hyaluronate plus hyaluronate knee injection (Experimental): oral hyaluronate plus hyaluronate knee injection
  Interventions: Drug: oral hyaluronate and injection
- hyaluronate knee injection (Placebo Comparator): hyaluronate knee injection
  Interventions: Drug: hyaluronate injection

INTERVENTIONS:
Drug: oral hyaluronate and injection — The patient receives oral hyaluronate and hyaluronate injection
  Arms: oral hyaluronate plus hyaluronate knee injection
Drug: hyaluronate injection — The patient receives hyaluronate injection only
  Arms: hyaluronate knee injection

SUMMARY:
The goal of this clinical trial is to investigate the effect of oral hyaluronate in patients with knee osteoarthritis. The main question it aims to answer is: the therapeutic effect in the combined treatment of oral nutritional supplement based on hyaluronic acid with hyaluronic acid intra-articular Injection on symptomatic knee osteoarthritis. Researchers will compare it to those who receive only hyaluronic acid injection to see if the combined treatment is better.

Participants will receive a total of three months of oral hyaluronate or placebo agents.

ELIGIBILITY:
Inclusion Criteria:

1. Radiological evidence of osteoarthritis Ahlbäck stage I-III.
2. Had knee effusion at the suprapatellar recess under ultrasonographic examination.
3. Age between 60 and 75 years old.

Exclusion Criteria:

1. Rheumatological disorders
2. Accidental trauma or fractures involving knees in the past three months
3. Neuropathic pain involving lower limbs
4. Central nervous system disorders including stroke, Parkinsonism, and spinal cord disorders.
5. Depression and cognitive problems
6. Pregnancy

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | From enrollment to the end of treatment at 12 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) aim to reveal pain, stiffness and function of the knee, the minimum and maximum values are 0 and 68, and a higher score mean a worse outcome.

SECONDARY OUTCOMES:
knee strength | From enrollment to the end of treatment at 12 weeks
  knee extension and flexion torque detected by isokinetic machine
Timed up and go test | From enrollment to the end of treatment at 12 weeks
  the time needed for a patient sits on a chair, stands up walks for 3 meters, and then go back down

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The patients we recruited are not willing to share their individual data

REFERENCES:
- [Background] Nelson FR, Zvirbulis RA, Zonca B, Li KW, Turner SM, Pasierb M, Wilton P, Martinez-Puig D, Wu W. The effects of an oral preparation containing hyaluronic acid (Oralvisc(R)) on obese knee osteoarthritis patients determined by pain, function, bradykinin, leptin, inflammatory cytokines, and heavy water analyses. Rheumatol Int. 2015 Jan;35(1):43-52. doi: 10.1007/s00296-014-3047-6. Epub 2014 Jun 5. PMID 24899570